CLINICAL TRIAL: NCT06056141
Title: Induction of Labour at Term With Low Dose Oral Misoprostol Versus a Foley Catheter: a Multicentre Randomised Controlled Trial
Brief Title: Induction of Labour at Term With Low Dose Oral Misoprostol Versus a Foley Catheter
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kazakhstan's Medical University "KSPH" (Other)
Collaborators: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Dilfuza Sultanmuratova, principal investigator, Kazakhstan's Medical University "KSPH"
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-23-2023
Record Dates: First submitted 2023-09-18; First posted 2023-09-28 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Induction of Labor
Keywords: Induction of labor; low dose misoprostol; Foley Catheter
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: multicentre randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Drug: Misoprostol 25mcg (200 mcg dissolved with 200 ml water and divided to 8 doses) every 2 hours
  Interventions: Drug: Misoprostol 200mcg Tab
- Group B (Active Comparator): Device: Foley Catheter Transcervical Foley catheter (silicone, size 20F with 30ml balloon)
  Interventions: Device: Foley Catheter

INTERVENTIONS:
Drug: Misoprostol 200mcg Tab — Misoprostol 200 mcg dissolvedwith 200 ml water and divided to 25ml solution every 2 hours per os for maximum of 8 doses
  Arms: Group A
Device: Foley Catheter — Transcervical Foley catheter (silicone, size 20F with 30ml balloon)
  Arms: Group B

SUMMARY:
Comparison of efficacy and safety of low-dose oral Misoprostol versus folley catheter for preinduction in women with an immature cervix at term.

DETAILED DESCRIPTION:
Open-label randomised trial in 2 hospitals in the Almaty,Kazakhstan. Women with a term singleton pregnancy in cephalic presentation, an unfavourable cervix, intact membranes, and without a previous caesarean section will be randomly allocated to 2 groups: 1 group -cervical ripening with 25 μg oral misoprostol once every 2 hour, 2 nd group- a 30 mL transcervical Foley catheter. The primary outcome will be vaginal delivery within 24 hours(to evaluate effectiveness) and secondary outcoms 1-5-min Apgar score and hospitalization in ICU, hyperstimulation frequency and hemorrage (for evaluating safety)

ELIGIBILITY:
Inclusion Criteria:

* women with an unfavourable cervix who will scheduled for induction of labour

Exclusion Criteria:

* Women with previous caesarean sections unable to give informed consent Multiple pregnancy History of allergy to misoprostol Ruptured membranes Chorioamnionitis All cases when physiological childbirth is impossible (placenta previa,transverse position of the fetus )

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Efficiency of induction | 24 hours.
  Number of Participants with vaginal births within 24 hours.

SECONDARY OUTCOMES:
Safety for baby | 5 min
  Rate of cases Apgar score <7 points
Safety for mother | during the labour induction
  incidence of hyperstimulation

CONTACTS AND LOCATIONS:
Locations (2):
- Kazakhstan (2):
  - City Perinatology Centre 3, Almaty
  - Center for Perinatology and Pediatric Cardiac Surgery, Almaty